CLINICAL TRIAL: NCT02663336
Title: Prevalence of Masked Hypertension in Nephrological Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Waid City Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: WaidBP16
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Masked Hypertension
Keywords: masked hypertension, chronic kidney disease
MeSH Terms: conditions — Masked Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CKD patients: Patients with chronic kidney disease, with diagnosed arterial hypertension and normal blood pressure during office blood pressure measurement. Comparison of ambulatory blood pressure (ABPM) with office blood pressure measurements (OBPM).
  Interventions: Other: Comparison ABPM with OBPM

INTERVENTIONS:
Other: Comparison ABPM with OBPM — No interventions

SUMMARY:
The purpose of this study is to determine the percentage of patients with masked hypertension in a population with chronic kidney disease. The investigators goal is to register prospectively ambulatory blood pressure measurement results of patients of a nephrological outpatient clinic with normal office blood pressure to finally find the percentage of masked hypertension in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-90 years
* Known arterial hypertension and antihypertensive medical treatment
* Office blood pressure < 140 mmHg systolic and <90 mmHg diastolic

Exclusion Criteria:

* Age <20 or >90 years

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease of the nephrological outpatient clinic of Waidspital with normal office blood pressure in the context of diagnosed arterial hypertension with or without antihypertensive medication
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2023-01 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with uncontrolled masked hypertension assessed by comparison of ambulatory blood pressure with office blood pressure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schleich, Principal Investigator — Stadtspital Waid Zurich Switzerland
Locations (1):
- Stadtspital Waid Zurich, Zurich, Switzerland